CLINICAL TRIAL: NCT06092489
Title: The Effectiveness of Graded Motor Imagery Therapy Applied in Addition to the Traditional Physiotherapy Program in Chronic Rotator Cuff-related Shoulder Pain.
Brief Title: Chronic Rotator Cuff-related Shoulder Pain and Graded Motor Imagery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuray Alaca (Other)
Responsible Party: Sponsor-Investigator, Nuray Alaca, Assoc, Prof. Nuray Alaca, Head of department Physiotherapy and Rehabilitation, Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/21-13
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain; Shoulder Pain
Keywords: chronic pain; shoulder pain; graded motor imagery
MeSH Terms: conditions — Chronic Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physiotherapy Program (Active Comparator): Self-stretching will encapsulate the upper trapezius, pectoralis minor, posterior. Each stretch will consist of 3 repetitions of 30 seconds with a 30 second break between repetitions. Strengthening exercises will be performed using elastic resistance bands (Theraband ®) with 4 levels of resistance (red, green, blue and grey). Sets can be easily changed (without the person reporting muscle fatigue) and progressed with resistance. The therapist will ask about the level of effort required for exercise exercises and whether it would be possible to increase the resistance level. The exercise consists of three sets of 10 repetitions and is completed with 1 rest between them. Strengthening exercises will include prone extension, prone external rotation with abduction, side lying external rotation and serratus anterior strengthening . These workouts and workouts are also arranged regularly. After exercise, ice will be applied to the shoulder for 15 minutes.
  Interventions: Other: traditional physiotherapy method
- Traditional Physiotherapy Program and Graded Motor Imagery Therapy (Experimental): The three different treatment techniques include left/right discrimination training, explicit motor imagery exercises and mirror therapy. These techniques are delivered sequentially but require a flexible approach from the patient and clinician to move forwards, backward and sideways in the treatment process to suit the individual. With patience, persistence and often lots of hard work, GMI gives new hope for treatment outcomes.
  Interventions: Other: graded motor imagery; Other: traditional physiotherapy method

INTERVENTIONS:
Other: graded motor imagery — The three different treatment techniques include left/right discrimination training, explicit motor imagery exercises and mirror therapy. These techniques are delivered sequentially but require a flexible approach from the patient and clinician to move forwards, backward and sideways in the treatment process to suit the individual. With patience, persistence and often lots of hard work, GMI gives new hope for treatment outcomes.
  Arms: Traditional Physiotherapy Program and Graded Motor Imagery Therapy
Other: traditional physiotherapy method — This protocol included stretching and strengthening exercises. Self-stretching will encapsulate the upper trapezius, pectoralis minor, posterior. Each stretch will consist of 3 repetitions of 30 seconds with a 30 second break between repetitions. Strengthening exercises will be performed using elastic resistance bands (Theraband ®) with 4 levels of resistance (red, green, blue and grey). Sets can be easily changed (without the person reporting muscle fatigue) and progressed with resistance. The therapist will ask about the level of effort required for exercise exercises and whether it would be possible to increase the resistance level. The exercise consists of three sets of 10 repetitions and is completed with 1 rest between them. Strengthening exercises will include prone extension, prone external rotation with abduction, side lying external rotation and serratus anterior strengthening.

SUMMARY:
Graded motor imagery (GMI) clinical conditions accompanied by many pain and movement problems; It is a treatment, education and rehabilitation process that is based on recently obtained scientific data and current clinical studies, is individually adapted and approaches the individual holistically with a biopsychosocial model. Nowadays, it is frequently used in the treatment of some neurological diseases. In addition, these approaches are also used in the treatment of some orthopedic diseases including chronic pain. There are a limited number of studies in which the mentioned approaches are used together in stages, and the stages are mostly used alone. Despite these positive results in favor of GMI, the fact that there is no study using the entire GMI treatment in chronic shoulder pain shows us that a randomized controlled and blinded study with high evidence value should be conducted on this subject. In addition, determining the effect of GMI on changes such as fear of pain, two-point discrimination, and left/right lateralization speed and accuracy task will help fill the literature gaps on this subject. In the light of this information, the question of planned master's thesis study is the effect of GMI treatment applied in addition to traditional physiotherapy in chronic rotator cuff-related shoulder pain on pain level, joint range of motion, functionality, pain-related fear, two-point discrimination and left/right lateralization speed and accuracy compared to only traditional physiotherapy. whether it is superior or not.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years Participants were classified with chronic Chronic Rotator Cuff-related Shoulder Pain if duration was equal or greater than 6 months, as recommended by the International Association for the Study of Pain for research purposes Pain at rest maximum 2 out of 10 on verbal numerical rating scale Pain over the deltoid and/or upper arm region for more than 4 weeks, pain associated with arm movement, and familiar pain reproduced with loading or resisted testing during abduction or external rotation of the arm Patient had to test positive at least 3 out of 5 symptoms-provoking tests: pain during Neer test, Hawkins-Kennedy test, Jobe test, painful arc between 60° and 120°, pain or weakness during external rotation resistance test

Exclusion Criteria:

Bilateral shoulder pain Corticosteroid injections less than 6 weeks prior to the enrolment Participants who were pregnant, Mini Mental State Examination score >24 Clinical signs of full-thickness rotator cuff tears (positive external and internal rotation lag tests or drop arm test) Evidence of adhesive capsulitis (50% or more than 30° loss of passive external rotation) Previous cervical, thoracic or shoulder surgery; recent fractures or dislocations on the painful shoulder Symptoms of cervical radiculopathy as primary complaint (tingling, radiating pain in the arm associated with neck complaints) Primary diagnosis of acromioclavicular pathology, shoulder instability Previous medical imaging confirming full-thickness rotator cuff tears or calcifications larger than 5mm Patients with competing pathologies (inflammatory arthritis, neurological disorders, fibromyalgia, malignancy) History of cancer, neurologic, systemic, rheumatic or vascular disorder and use of psychiatric medication Participants performing overhead sport activities for more than 4hours/week

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NPRS-11) | Change from baseline range of motion at 6th week
  he Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain).0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
The Shoulder Pain and Disability Index | Change from baseline score of The Shoulder Pain and Disability Index at 6th week
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability between 0 to 100, with a higher value indicating worse condition.
Global Rating of Change scale | Change from baseline Global Rating of Change scale at 6th week
  Patient satisfaction regarding improvement in shoulder function will be evaluated by the Global Rating of Change scale. All participants will be asked to rate their condition after a six-week intervention period compared to baseline by indicating whether they have improved significantly, improved slightly, unchanged, deteriorated slightly, or deteriorated significantly between -3 to +3, with a higher value indicating better condition in this study.
Central Sensitization Scale | Change from baseline score of Central Sensitization Scale scale at 6th week
  Central Sensitization Scale, which can be applied in the presence of chronic pain, is used in central sensitization syndromes. It consists of two parts. Part A of the scale includes a Likert scale (0-4 points) that questions health-related symptoms. This section is scored from 0 to 100, with higher numbers being associated with a higher degree of central sensitization. Scores of 40 and above indicate the presence of central sensitization. In section B, it questions whether any of the central sensitization syndromes have been diagnosed before.

SECONDARY OUTCOMES:
Range of motion | Change from baseline range of motion at 6th week]
  Shoulder range of motion is the capability of a joint to go through its complete spectrum of movements.
Pressure Pain Threshold | Change from baseline Pressure Pain Threshold at 6th week
  A digital pressure algometer will be applied to the web space of the foot opposite the trigger point. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold).
Pain Catastrophizing Scale | Change from baseline score of Pain Catastrophizing Scale at 6th week
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain.The person may score a total of 52 (Pain Catastrophizing Scale). A high score indicates a high level of catastrophic.
Fear avoidance belief questionnaire (FABQ) | Change from baseline score of Fear avoidance belief questionnaire at 6th week
  Fear avoidance belief questionnaire FABQ) is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)
The two-point discrimination test | Change from baseline two-point discrimination at 6th week
  The two-point discrimination test is used to assess if the patient is able to identify two close points on a small area of skin, and how fine the ability to discriminate this are. It is a measure of tactile agnosia, or the inability to recognize these two points despite intact cutaneous sensation and proprioception
Left/right discrimination (Lateralization) | Change from baseline Left/right discrimination at 6th week
  Right-Left Discrimination will be evaluated with Recognise™ applications (Shoulder and Hand) developed by the "Neuro Orthopedic Institute".
Kinesthetic and Visual Imagery Questionnaire (KVIQ) | Change from baseline Kinesthetic and Visual Imagery Questionnaire at 6th week
  Motor imagery ability will be assessed with the Kinesthetic and Visual Imagery Questionnaire (KVIQ). The participant gives a score between 1 and 5 for the image he/she imagines: "1 point: no image, 5 points: as clear as the original." This process is repeated for each task and at the end of the survey, kinesthetic imagery score, visual imagery score and total score are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray ALACA, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sirlan S, Alaca N, Yarar HA, Basci O. Graded motor imagery as an adjunct to comprehensive physiotherapy in chronic rotator cuff-related pain: a single blind randomized controlled trial. BMC Musculoskelet Disord. 2025 Jul 3;26(1):588. doi: 10.1186/s12891-025-08783-w. PMID 40611093